CLINICAL TRIAL: NCT00114569
Title: Use of Lorazepam for the Treatment of Status Epilepticus
Brief Title: Lorazepam for the Treatment of Status Epilepticus in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: James Chamberlain, Children's National Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHSN275200403393C; HHSN275200403393C
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2009-05

CONDITIONS: Status Epilepticus
Keywords: children; status epilepticus; lorazepam; safety; pharmacokinetics; status epilepticus in children
MeSH Terms: conditions — Status Epilepticus | interventions — Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lorazepam

SUMMARY:
The purpose of this study is to gather the data to: 1) determine the best dose, and 2) evaluate its effectiveness and safety in stopping seizures. Part 1 is a pharmacokinetic study (study of how much drug is found in the body after it is given through a vein and how fast the body gets rid of the drug).

DETAILED DESCRIPTION:
Lorazepam is in a class of drugs called benzodiazepines that is used to treat seizures. Lorazepam has been widely used to treat children who have repeated or long seizures, a condition known as status epilepticus (SE). However, lorazepam is not currently approved by the FDA for use in children under 18 years of age. Therefore, the purpose of this study is to gather the data needed for FDA approval. Specifically, we will 1) determine the best dose, and 2) evaluate its effectiveness and safety in stopping seizures. Part 1 is a pharmacokinetic study. These are studies designed to identify and describe one or more of the following basic pharmacological concepts in humans: absorption (i.e. how much gets into the body); distribution (i.e. where it goes in the body); and metabolism and elimination (i.e. how the body gets rid of the medication and how long it takes). The study procedures involve taking blood samples from children, taking their vital signs, and conducting physical examinations. Informed consent will be obtained from all participants as required by federal guidelines. Patients will be divided into two groups. The first group will be patients who present to one of the 10 participating Emergency Rooms (ERs) in status epilepticus (repeated or continuous seizures). We will either ask for consent in the ER, or if we know they have a seizure disorder and have frequent visits to the ER, consent them beforehand for future visits to the ER. The second group will include patients who have a known seizure disorder and agree to be electively admitted to the hospital for a dose of lorazepam when they are not having seizures. We will draw blood samples from patients for up to 48 hours and then follow up via telephone for 30 days from the day the medication was given to assess for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Generalized tonic clonic seizures within 1 hour OR 2 or more generalized tonic clonic seizures in rapid succession with no recovery of consciousness between seizures OR a single ongoing generalized tonic clonic seizure which has lasted at least 5 minutes

Exclusion Criteria:

* Inability to obtain informed consent or assent
* Sustained hypotension
* Significant arrhythmia
* Known hypersensitivity to or contraindication to use of benzodiazepines
* Use of lorazepam within 4 days of study drug dosing
* American Association of Anesthesiology (ASA) Class > 1

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2005-03; Primary Completion 2007-04 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacokinetics of two different doses (0.05 and 0.1 mg/kg) IV lorazepam

SECONDARY OUTCOMES:
safety of IV lorazepam

CONTACTS AND LOCATIONS:
Overall Officials: James Chamberlain, MD, Principal Investigator — Children's National Medical Center, Washington, D.C.
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States